CLINICAL TRIAL: NCT02106351
Title: A Phase III, Multicentre, Double Blind, Prospective, Randomised, Controlled, Multiple Treatment Study Assessing Efficacy And Safety Of DYSPORT® Used In The Treatment Of Upper Limb Spasticity In Children
Brief Title: Efficacy And Safety Of Dysport In The Treatment Of Upper Limb Spasticity In Children
Acronym: PUL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Y-52-52120-153; 2010-021817-22 (EudraCT Number)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Results first posted 2019-12-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Upper Limb Spasticity (Altered Skeletal Muscle Performance) in Children
MeSH Terms: interventions — Botulinum Toxins, Type A; abobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Group A - Treatments 1, 2, 3 and 4: Dysport 16 Units (U)/kg in one upper extremity (the study limb).
  Interventions: Biological: Botulinum toxin type A
- Group B (Experimental): Group B - Treatments 1, 2, 3 and 4: Dysport 8 U/kg in one upper extremity (the study limb).
  Interventions: Biological: Botulinum toxin type A
- Group C (Experimental): Group C - Treatment 1: Dysport 2 U/kg in one upper extremity (the study limb).
  Group C - Treatments 2, 3 and 4: Dysport 8 or 16 U/kg in one upper extremity (the study limb).
  Interventions: Biological: Botulinum toxin type A

INTERVENTIONS:
Biological: Botulinum toxin type A — Subjects randomised to receive Dysport 2 U/kg, 8 U/kg or 16 U/kg administered intramuscularly in the study limb.
  Other Names: AbobotulinumtoxinA (Dysport®)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of multiple doses of Dysport used in the treatment of upper limb spasticity (altered skeletal muscle performance) in children with cerebral palsy (CP).

ELIGIBILITY:
Inclusion Criteria:

* Upper limb spasticity due to cerebral palsy
* Body weight 10 kg or over
* MAS score of 2 or more in affected elbow or wrist flexors

Exclusion Criteria:

* Fixed myocontracture
* Previous phenol or alcohol injection within 1 year
* Severe athetoid or dystonic movements
* Previous or planned surgery for spasticity in elbow or wrist flexors
* Neuromuscular disorders
* Previous Rhizotomy within 6 months
* Intrathecal baclofen within 30 days

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 212 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-09-21 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (31):
- United States (12):
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - New Orleans, Louisiana
  - Royal Oak, Michigan
  - Saint Paul, Minnesota
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - New York, New York
  - Columbus, Ohio
  - Portland, Oregon
  - Austin, Texas
  - Dallas, Texas
- Brussels, Belgium
- Czechia (2):
  - Brno
  - Prague
- Israel (5):
  - Beersheba
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
  - Tel Litwinsky
- Mexico (3):
  - La Paz, Baja California Sur
  - Celaya
  - Monterrey
- Poland (3):
  - Gdansk
  - Poznan
  - Wiązowna
- Spain (2):
  - Barcelona
  - Terrassa
- Turkey (Türkiye) (3):
  - Istanbul
  - Izmir
  - Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized, and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers

REFERENCES:
- [Derived] Delgado MR, Tilton A, Carranza-Del Rio J, Dursun N, Bonikowski M, Aydin R, Maciag-Tymecka I, Oleszek J, Dabrowski E, Grandoulier AS, Picaut P; Dysport in PUL study group. Efficacy and safety of abobotulinumtoxinA for upper limb spasticity in children with cerebral palsy: a randomized repeat-treatment study. Dev Med Child Neurol. 2021 May;63(5):592-600. doi: 10.1111/dmcn.14733. Epub 2020 Nov 18. PMID 33206382
- [Derived] Shierk A, Jimenez-Moreno AC, Roberts H, Ackerman-Laufer S, Backer G, Bard-Pondarre R, Cekmece C, Pyrzanowska W, Vilain C, Delgado MR. Development of a Pediatric Goal-Centered Upper Limb Spasticity Home Exercise Therapy Program for Use in a Phase-III Trial of Abobotulinumtoxina (Dysport(R)). Phys Occup Ther Pediatr. 2019;39(2):124-135. doi: 10.1080/01942638.2018.1486346. Epub 2018 Sep 11. PMID 30204515

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female subjects aged between 2 and 17 years with upper limb spasticity due to cerebral palsy (CP) were recruited from April 2014 and the study completed in September 2018. Subjects could receive a maximum of 4 treatment cycles (TC) over a minimum of 1 year and maximum of 1 year and 9 months, with at least 16 weeks between each TC.
Pre-assignment Details: Subjects had a body weight ≥10 kilograms (kg), increased muscle tone/spasticity in at least 1 upper limb, a modified Ashworth scale (MAS) score ≥2 in the upper limb primary targeted muscle group (PTMG) of the study limb at baseline. Subjects were stratified according to age (2-9 and 10-17 years) and Botulinum Toxin (BTX) naïve or non-naïve status.
Groups:
- Dysport 2 U/kg: Subjects were randomised to receive Dysport 2 Units per kg (U/kg) by intramuscular (IM) injection into the study upper limb in TC 1 and Dysport 8 U/kg or 16 U/kg in subsequent TCs (2, 3 and 4). Retreatment was based on clinical need with a minimum retreatment interval of 16 weeks. In all TCs the dose was divided between the PTMG (elbow or wrist flexors) and a number of other upper limb muscles based on clinical presentation. From TC 2 onwards dose adaptation was permitted as well as treatment of the non-study upper limb and lower limbs.
- Dysport 8 U/kg: Subjects were randomised to receive Dysport 8 U/kg by IM injection into the study upper limb in TC 1 and all subsequent TCs (2, 3 and 4), up to a maximum of 320 U. Retreatment was based on clinical need with a minimum retreatment interval of 16 weeks. In all TCs the dose was divided between the PTMG (elbow or wrist flexors) and a number of other upper limb muscles based on clinical presentation. From TC 2 onwards dose adaptation was permitted as well as treatment of the non-study upper limb and lower limbs.
- Dysport 16 U/kg: Subjects were randomised to receive Dysport 16 U/kg by IM injection into the study upper limb in TC 1 and all subsequent TCs (2, 3 and 4), up to a maximum of 640 U. Retreatment was based on clinical need with a minimum retreatment interval of 16 weeks. In all TCs the dose was divided between the PTMG (elbow or wrist flexors) and a number of other upper limb muscles based on clinical presentation. From TC 2 onwards dose adaptation was permitted as well as treatment of the non-study upper limb and lower limbs.
Period: Treatment Cycle 1
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Started | 71 | 70 | 71
Received Treatment in TC 1 | 70 | 70 | 70
Completed | 66 | 67 | 67
Not Completed | 5 | 3 | 4
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Consent withdrawn | 1 | 0 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Other | 0 | 3 | 1
Not completed — Randomised but not treated | 1 | 0 | 1
Period: Treatment Cycle 2
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Started | 0 (Subjects who received Dysport 2 U/kg in TC 1 were randomised to receive 8 or 16 U/kg in TCs 2-4.) | 88 (Not all subjects who completed TC 1 required retreatment in TC 2.) | 90 (Not all subjects who completed TC 1 required retreatment in TC 2.)
Completed | 0 | 83 | 87
Not Completed | 0 | 5 | 3
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Consent withdrawn | 0 | 1 | 1
Not completed — Other | 0 | 2 | 2
Period: Treatment Cycle 3
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Started | 0 | 49 (Not all subjects who completed TC 2 required retreatment in TC 3.) | 58 (Not all subjects who completed TC 2 required retreatment in TC 3.)
Completed | 0 | 45 | 53
Not Completed | 0 | 4 | 5
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Consent withdrawn | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 0 | 2 | 3
Period: Treatment Cycle 4
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Started | 0 | 22 (Not all subjects who completed TC 3 required retreatment in TC 4.) | 33 (Not all subjects who completed TC 3 required retreatment in TC 4.)
Completed | 0 | 21 | 31
Not Completed | 0 | 1 | 2
Not completed — Consent withdrawn | 0 | 0 | 2
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are presented for the safety population, which consisted of all randomised subjects who received at least 1 injection of the study treatment.
Groups:
- Dysport 2 U/kg: Subjects were randomised to receive Dysport 2 U/kg by IM injection into the study upper limb in TC 1 and Dysport 8 U/kg or 16 U/kg in subsequent TCs (2, 3 and 4).
- Dysport 8 U/kg: Subjects were randomised to receive Dysport 8 U/kg by IM injection into the study upper limb in TC 1 and all subsequent TCs (2, 3 and 4), up to a maximum of 320 U.
- Dysport 16 U/kg: Subjects were randomised to receive Dysport 16 U/kg by IM injection into the study upper limb in TC 1 and all subsequent TCs (2, 3 and 4), up to a maximum of 640 U.
- Total: Total of all reporting groups
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg | Total
Number analyzed (Participants) | 70 | 70 | 70 | 210
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.91 (4.55) | 8.97 (4.27) | 9.17 (4.30) | 9.02 (4.36)
Age, Customized [Count of Participants; unit: Participants]
  2 - 9 Years | 40 | 40 | 40 | 120
  10 - 17 Years | 30 | 30 | 30 | 90
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 24 | 28 | 84
  Male | 38 | 46 | 42 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 0 | 3
  Black or African American | 7 | 6 | 3 | 16
  White | 49 | 54 | 54 | 157
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Multiple | 12 | 8 | 13 | 33
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 13 | 15 | 44
  Not Hispanic or Latino | 54 | 57 | 55 | 166
BTX Status [Count of Participants; unit: Participants]
  BTX naïve | 25 | 23 | 24 | 72
  BTX non-naïve | 45 | 47 | 46 | 138
Baseline MAS Score in the PTMG [Mean (Standard Deviation); unit: score on a scale] — The MAS has 6 grades ranging from 0 to 4 with higher scores indicate greater muscle tone. Where, 0 = no increase in muscle tone, 1 = slight increase in muscle tone, manifested by a catch + release or minimal resistance at end of range of motion (ROM), 1+ = slight increase in muscle tone, manifested by a catch and then minimal resistance throughout remainder (less than half) of ROM, 2 = more marked increase in muscle tone, 3 = considerable increase in muscle tone and 4 = affected part(s) rigid in flexion/extension. '1+' was given a derived score of '2'; following scores were incremented by 1.
  score on a scale | 3.1 (0.3) | 3.1 (0.3) | 3.1 (0.5) | 3.1 (0.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to TC 1, Week 6 in MAS Score in the TC 1 PTMG
Description: The MAS was used to assess muscle tone in the upper limb PTMG and consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM) when the affected part is moved in flexion or extension, 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension). The original score '+1' was given a derived numeric score of '2' and the higher numeric scores were incremented by 1 so that the MAS score range was from 0 to 5 with higher scores indicating greater muscle tone. A negative change from baseline indicates a decrease in muscle tone.
Time Frame: Baseline (TC 1, Day 1) and TC 1, Week 6.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
score on a scale | -1.5 (1.1) | -1.9 (1.0) | -2.2 (0.9)
Statistical Analysis 1: Comparison: Dysport 2 U/kg vs Dysport 8 U/kg; The treatment difference between Dysport 8 U/kg and Dysport 2 U/kg was analysed using an analysis of covariance (ANCOVA) on the ranked changes from baseline. The model included treatment group, the baseline value, the 2 stratification factors (age range and BTX status at baseline) and the pooled centre as fixed effects. The derived least squares (LS) means were back transformed to the original scale and the treatment difference determined; Test type: Superiority; p = 0.0118, ANCOVA — The 2-tailed significance level was 0.05; ANCOVA is performed on the ranked values; LS mean difference back transformed = -0.4
Statistical Analysis 2: Comparison: Dysport 2 U/kg vs Dysport 16 U/kg; The treatment difference between Dysport 16 U/kg and Dysport 2 U/kg was analysed using an ANCOVA on the ranked changes from baseline. The model included treatment group, the baseline value, the 2 stratification factors (age range and BTX status at baseline) and the pooled centre as fixed effects. The derived LS means were back transformed to the original scale and the treatment difference determined; Test type: Superiority; p < 0.0001, ANCOVA — The 2-tailed significance level was 0.05; ANCOVA is performed on the ranked values; LS mean difference back transformed = -0.7

2. Secondary Outcome: Mean Physician's Global Assessment (PGA) Score at TC 1, Week 6
Description: The PGA of treatment response was assessed by asking the investigator the following question: 'How would you rate the response to treatment in the subject's upper limb since the start of the study?'. Answers were on a 9-point rating scale (-4: markedly worse, -3: much worse, -2: worse, -1: slightly worse, 0: no change, +1: slightly improved, +2: improved, +3: much improved and +4: markedly improved). The mean scores for each treatment group at TC 1, Week 6 are presented.
Time Frame: TC 1, Week 6.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects with data available are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 68 | 69 | 70
score on a scale | 1.7 (0.9) | 2.0 (0.9) | 2.0 (0.9)
Statistical Analysis 1: Comparison: Dysport 2 U/kg vs Dysport 8 U/kg; The treatment difference between Dysport 8 U/kg and Dysport 2 U/kg was analysed using an analysis of variance (ANOVA) on the rank of the PGA score at TC 1, Week 6. The model included treatment group, the 2 stratification factors (age range and BTX status at baseline) and the centre as fixed effects. The derived LS means were back transformed to the original scale and the treatment difference determined; Test type: Superiority; p = 0.2043, ANOVA — The two-tailed significance level was 0.05; ANOVA was performed on ranked values; LS mean difference back transformed = 0.2
Statistical Analysis 2: Comparison: Dysport 2 U/kg vs Dysport 16 U/kg; The treatment difference between Dysport 16 U/kg and Dysport 2 U/kg was analysed using an ANOVA on the rank of the PGA score at TC 1, Week 6. The model included treatment group, the 2 stratification factors (age range and BTX status at baseline) and the centre as fixed effects. The derived LS means were back transformed to the original scale and the treatment difference determined; Test type: Superiority; p = 0.1880, ANOVA — The two-tailed significance level was 0.05; ANOVA was performed on ranked values; LS mean difference back transformed = 0.2

3. Secondary Outcome: Mean Goal Attainment Scale (GAS) Total Score at TC 1, Week 6
Description: The GAS is a functional 5-point scale used to measure progress towards individual therapy goals. At start of each TC, 1 to 3 individual goals were defined for each subject by investigator and child's parents/guardians/caregivers prior to treatment. Outcome to reach each goal was rated on a 5-point scale ranging from -2 to +2 (-2: much less than expected outcome, -1: somewhat less than expected outcome, 0: expected outcome, +1: somewhat more than expected outcome, +2: much more than expected outcome). Higher score indicates a better outcome. A GAS T-score was calculated as: 50+(10∑_(i=1)^n wi xi)/√(0.7∑_(i=1)^n wi^2 +0.3(∑_(i=1)^n wi)^2) where, xi = rating of ith goal post-baseline; wi = weight of ith goal, calculated as importance * difficulty as defined at baseline; n = number of goals assessed at baseline and post-baseline. A GAS T-score of 50 indicates goals achieved as expected. Scores below 50 reflect under attainment of goals and scores above 50 reflect over attainment of goals.
Time Frame: TC 1, Week 6.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 68 | 66 | 70
T-score | 51.3 (9.9) | 52.6 (10.1) | 52.0 (9.6)
Statistical Analysis 1: Comparison: Dysport 2 U/kg vs Dysport 8 U/kg; The treatment difference between Dysport 8 U/kg and Dysport 2 U/kg was analysed using ANOVA on the GAS Total score at TC 1, Week 6. The model included treatment group, the 2 stratification factors (age range and BTX status at baseline) and the centre as fixed effects; Test type: Superiority; p = 0.7648, ANOVA — The two-tailed significance level was 0.05; LS mean difference = 0.5, 95% CI 2-sided [-2.7 to 3.7]
Statistical Analysis 2: Comparison: Dysport 2 U/kg vs Dysport 16 U/kg; The treatment difference between Dysport 16 U/kg and Dysport 2 U/kg was analysed using ANOVA on the GAS Total score at TC 1, Week 6. The model included treatment group, the 2 stratification factors (age range and BTX status at baseline) and the centre as fixed effects; Test type: Superiority; p = 0.7429, ANOVA — The two-tailed significance level was 0.05; LS mean difference = 0.5, 95% CI 2-sided [-2.6 to 3.7]

4. Other Pre Specified Outcome: Mean Change From Baseline to TC 1 Week 16 in MAS Score in the TC 1 PTMG
Description: as for outcome 1
Time Frame: Baseline (TC 1, Day 1) and TC 1, Week 16.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects with data available at the timepoint analysed are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 68 | 68 | 68
score on a scale | -1.0 (1.0) | -1.4 (1.1) | -1.6 (1.2)

5. Other Pre Specified Outcome: Mean Change From Baseline to TC 1 Weeks 6 and 16 in MAS Score in the Elbow Flexors of the Study Limb
Description: The MAS was used to assess muscle tone in the upper limb PTMG and consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM) when the affected part is moved in flexion or extension, 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension). The original score '+1' was given a derived numeric score of '2' and the higher numeric scores were incremented by 1 so that the MAS score range was from 0 to 5 with higher scores indicating greater muscle tone. A negative change from baseline indicates a decrease in muscle tone. Data is presented for subjects injected in the elbow flexors.
Time Frame: Baseline (TC 1, Day 1) and TC 1, Weeks 6 and 16.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects with data available at each timepoint and who were injected in the elbow flexors are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
score on a scale
  Week 6: number analyzed (Participants) | 63 | 63 | 62
  Week 6 | -1.0 (1.1) | -1.7 (1.1) | -1.9 (1.2)
  Week 16: number analyzed (Participants) | 62 | 62 | 60
  Week 16 | -0.6 (1.0) | -1.2 (1.2) | -1.3 (1.4)

6. Other Pre Specified Outcome: Mean Change From Baseline to TC 1 Weeks 6 and 16 in MAS Score in the Wrist Flexors of the Study Limb
Description: The MAS was used to assess muscle tone in the upper limb PTMG and consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM) when the affected part is moved in flexion or extension, 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension). The original score '+1' was given a derived numeric score of '2' and the higher numeric scores were incremented by 1 so that the MAS score range was from 0 to 5 with higher scores indicating greater muscle tone. A negative change from baseline indicates a decrease in muscle tone. Data is presented for subjects injected in the wrist flexors.
Time Frame: Baseline (TC 1, Day 1) and TC 1, Weeks 6 and 16.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects with data available at each timepoint and who were injected in the wrist flexors are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
score on a scale
  Week 6: number analyzed (Participants) | 50 | 53 | 61
  Week 6 | -1.3 (1.1) | -1.5 (1.2) | -1.7 (1.3)
  Week 16: number analyzed (Participants) | 50 | 53 | 59
  Week 16 | -0.9 (1.2) | -1.0 (1.2) | -1.3 (1.2)

7. Other Pre Specified Outcome: Mean Change From Baseline to TC 1 Weeks 6 and 16 in MAS Score in the Finger Flexors of the Study Limb
Description: The MAS was used to assess muscle tone in the upper limb PTMG and consists of 6 grades: 0 (no increase in muscle tone), 1 (slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the ROM) when the affected part is moved in flexion or extension, 1+ (slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM), 2 (more marked increase in muscle tone), 3 (considerable increase in muscle tone) or 4 (affected part(s) rigid in flexion or extension). The original score '+1' was given a derived numeric score of '2' and the higher numeric scores were incremented by 1 so that the MAS score range was from 0 to 5 with higher scores indicating greater muscle tone. A negative change from baseline indicates a decrease in muscle tone. Data is presented for subjects injected in the finger flexors.
Time Frame: Baseline (TC 1, Day 1) and TC 1, Weeks 6 and 16.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects with data available at each timepoint and who were injected in the finger flexors are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
score on a scale
  Week 6: number analyzed (Participants) | 23 | 23 | 19
  Week 6 | -0.8 (0.9) | -1.8 (1.1) | -1.9 (1.0)
  Week 16: number analyzed (Participants) | 22 | 23 | 19
  Week 16 | -0.8 (1.3) | -1.3 (0.8) | -1.8 (1.0)

8. Other Pre Specified Outcome: Mean PGA Score at TC 1 Week 16
Description: The PGA of treatment response was assessed by asking the investigator the following question: 'How would you rate the response to treatment in the subject's upper limb since the start of the study?'. Answers were on a 9-point rating scale (-4: markedly worse, -3: much worse, -2: worse, -1: slightly worse, 0: no change, +1: slightly improved, +2: improved, +3: much improved and +4: markedly improved). The mean scores for each treatment group at TC 1 Week 16 are presented.
Time Frame: Baseline (TC 1, Day 1) and TC 1, Week 16.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects with available data at the timepoint analysed are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
score on a scale | 1.7 (1.0) | 1.6 (1.1) | 1.9 (1.2)

9. Other Pre Specified Outcome: Mean GAS Total Score at TC 1, Week 16
Description: as for outcome 3
Time Frame: Baseline (TC 1, Day 1) and TC 1, Week 16.
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
T-score | 54.7 (9.8) | 54.2 (9.7) | 55.1 (10.1)

10. Other Pre Specified Outcome: Mean Change From Baseline to TC 1, Week 16 in the Paediatric Quality of Life (PedsQL) Scores
Description: Parents/guardians completed questionnaires on their child's quality of life. The PedsQL parent inventory measured healthcare concepts for children/adolescents aged 2-18 years. The Generic Core Scales include physical, emotional, social and school aspects. The CP module was also completed. Scores were transformed on a scale from 0 to 100 with higher scores indicating a better quality of life. Mean changes from baseline to TC 1, Week 16 are presented for the General Core Scale and for the CP module. A positive change from baseline indicates an improvement in quality of life.
Time Frame: Baseline (TC 1, Day 1) and TC 1, Week 16.
Population: The mITT population consisted of all randomised subjects who received at least 1 injection of the study treatment and had a MAS score in the PTMG assessed at both baseline (TC 1, Day 1) and at TC 1, Week 6. Subjects who were assessed at each timepoint are presented.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dysport 2 U/kg | Dysport 8 U/kg | Dysport 16 U/kg
Number analyzed (Participants) | 69 | 69 | 70
score on a scale
  Generic Core Scale: number analyzed (Participants) | 67 | 67 | 67
  Generic Core Scale | 3.4 (9.7) | 3.4 (17.1) | 2.0 (12.0)
  CP Module: number analyzed (Participants) | 64 | 64 | 65
  CP Module | 4.8 (16.8) | 2.1 (14.9) | 2.8 (16.2)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from the first injection of study treatment up to the end of TC 4 (up to 21 months).
Description: TEAEs are reported for the dose received prior to onset of the AE. Due to dose adaption due to safety lower doses were permitted for TCs 2 - 4.
Groups:
- TC1: Dysport 2 U/kg: Subjects randomised to Dysport 2 U/kg in TC 1.
- TC 1: Dysport 8 U/kg: Subjects randomised to Dysport 8 U/kg in TC 1.
- TC 1: Dysport 16 U/kg: Subjects randomised to Dysport 16 U/kg in TC 1.
- TC 2: Dysport 8 U/kg: Subjects who received Dysport 8 U/kg in TC 2.
- TC 2: Dysport 16 U/kg: Subjects who received Dysport 16 U/kg in TC 2.
- TC 3: Dysport 8 U/kg: Subjects who received Dysport 8 U/kg in TC 3.
- TC 3: Dysport 16 U/kg: Subjects who received Dysport 16 U/kg in TC 3.
- TC 4: Dysport 8 U/kg: Subjects who received Dysport 8 U/kg in TC 4.
- TC 4: Dysport 16 U/kg: Subjects who received Dysport 16 U/kg in TC 4.
Arm/Group | TC1: Dysport 2 U/kg | TC 1: Dysport 8 U/kg | TC 1: Dysport 16 U/kg | TC 2: Dysport 8 U/kg | TC 2: Dysport 16 U/kg | TC 3: Dysport 8 U/kg | TC 3: Dysport 16 U/kg | TC 4: Dysport 8 U/kg | TC 4: Dysport 16 U/kg
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/70 | 0/70 | 0/88 | 0/90 | 0/49 | 0/58 | 0/22 | 0/33
Serious Adverse Events (participants affected / at risk) | 4/70 | 2/70 | 2/70 | 6/88 | 1/90 | 3/49 | 2/58 | 2/22 | 1/33
Other Adverse Events (participants affected / at risk) | 15/70 | 23/70 | 19/70 | 18/88 | 17/90 | 14/49 | 10/58 | 14/22 | 5/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TC1: Dysport 2 U/kg (N=70) | TC 1: Dysport 8 U/kg (N=70) | TC 1: Dysport 16 U/kg (N=70) | TC 2: Dysport 8 U/kg (N=88) | TC 2: Dysport 16 U/kg (N=90) | TC 3: Dysport 8 U/kg (N=49) | TC 3: Dysport 16 U/kg (N=58) | TC 4: Dysport 8 U/kg (N=22) | TC 4: Dysport 16 U/kg (N=33)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 | 0
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral ventricle dilatation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular malignant teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle release (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ostectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiotherapy to bone (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram ST segment elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scoliosis surgery (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TC1: Dysport 2 U/kg (N=70) | TC 1: Dysport 8 U/kg (N=70) | TC 1: Dysport 16 U/kg (N=70) | TC 2: Dysport 8 U/kg (N=88) | TC 2: Dysport 16 U/kg (N=90) | TC 3: Dysport 8 U/kg (N=49) | TC 3: Dysport 16 U/kg (N=58) | TC 4: Dysport 8 U/kg (N=22) | TC 4: Dysport 16 U/kg (N=33)
Viral upper respiratory tract infection (Infections and infestations) | 10 (13) | 6 (7) | 6 (7) | 7 (8) | 6 (6) | 6 (9) | 5 (8) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 5 (6) | 6 (8) | 8 (10) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 6 (8) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (5) | 2 (2) | 7 (8) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 4 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intenational normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-07-24): https://cdn.clinicaltrials.gov/large-docs/51/NCT02106351/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02106351/SAP_001.pdf